CLINICAL TRIAL: NCT05022004
Title: Therapeutic Equivalence Study of Generic Brinzolamide 1% Ophthalmic Suspension Compared to Reference Listed Drug Azopt® (Brinzolamide) Ophthalmic Suspension 1% in Subjects With Primary Open Angle Glaucoma or Ocular Hypertension.
Brief Title: A Therapeutic Equivalence Study in Subjects With Primary Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BRIN-20-01
Record Dates: First submitted 2021-08-19; First posted 2021-08-26 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-12

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BRIN-20-01 (Experimental)
  Interventions: Drug: Brinzolamide ophthalmic suspension
- Azopt® (Active Comparator)
  Interventions: Drug: Azopt®

INTERVENTIONS:
Drug: Brinzolamide ophthalmic suspension — dose: one drop of study medication; frequency: three times a day; route of administration: Topical ocular administration; duration of therapy: 6 weeks
  Arms: BRIN-20-01
Drug: Azopt® — dose: one drop of study medication; frequency: three times a day; route of administration: Topical ocular administration; duration of therapy: 6 weeks
  Arms: Azopt®

SUMMARY:
This is a randomized, Investigator-masked, multi-center, parallel group, therapeutic equivalence study with clinical endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Male or nonpregnant female aged 18 years or older with chronic open angle glaucoma or ocular hypertension in both eyes.
* Provide signed and dated informed consent in accordance with good clinical practice and local legislation prior to any study procedure.
* Be able and willing to follow study instructions and complete all required visits.
* Subject requires treatment of both eyes and is able to discontinue use of all ocular hypotensive medication(s) or switch ocular hypotensive medications and undergo appropriate washout period.

Exclusion Criteria:

* Subjects with angle closure glaucoma
* Females who are pregnant, breast feeding, or planning a pregnancy.
* Females of childbearing potential who do not agree to utilize an adequate form of contraception.
* Current, or past history of, severe hepatic or renal impairment
* Current, or history within 2 months prior to baseline of, significant ocular disease
* Functionally significant visual field loss
* Contraindication to brinzolamide or sulfonamide therapy or known hypersensitivity to any component of brinzolamide or sulfonamide therapy
* Subjects currently in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2023-01-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- India (14):
  - GMC, Srikakulam, Srikakulam, Andhra Pradesh
  - Dr. RSPR Govt Regional Eye Hospital; Vishakapatnam, Visakhapatnam, Andhra Pradesh
  - Rising Retina Clinic, Ahmedabad, Gujarat
  - Bhavna Super speciality Eye care, Surat, Gujarat
  - Dr. BR Ambedkar Medical College and hospital, Bangalore, Karnataka
  - Bhagwan Mahaveer Jain Hospital, Bangalore, Karnataka
  - KLE's Dr. Prabhakar Kore Hospital & Medical Research Center, Belagavi, Karnataka
  - K R Hospital, Mysore Medical College and Research Institute, Mysuru, Karnataka
  - Shanti Saroj Netralay, Miraj, Maharashtra
  - Omkar Eye Care Center, Mumbai, Maharashtra
  - Acharya Vinoba Bhave Rural Hospital, Jawaharlal Nehru Medical College, Datta Meghe Institute of Medical Sciences, Wardha, Maharashtra
  - Sankara Nethralaya, Chennai, Tamil Nadu
  - Dr Agarwal's Eye Hospital, Tirunelveli, Tamil Nadu
  - Heritage Institute of Medical Sciences, Varanasi, Uttar Pradesh
- Russia (26):
  - Institute of Human Brain of the Russian Academy of Science, 197376, Academ. Pavlov street 12 AP, StPetersburg, Russia, Saint Petersberg, Sankt-Peterburg
  - Republican clinical ophthalmological hospital of Ministry of Health of Republic of Tatarstan named after E.V. Adamyuk, Kazan', Tatarstan Republic
  - Federal State Autonomous Institution "Interdistrict Scientific and Technical Complex "Eye Microsurgery" named after Academician S.N. Fedorov" of the Ministry of Healthcare of the Russian Federation, Cheboksary
  - Healthcare Organization "Eye Center", Limited Liability Company, Chelyabinsk
  - Federal State Autonomous Institution "Interdistrict Scientific and Technical Complex "Eye Microsurgery" named after Academician S.N. Fedorov" of the Ministry of Healthcare of the Russian Federation, Irkutsk
  - Ivanovo Regional Clinical Hospital, Ivanovo
  - "Eye Microsurgery" n a Academician S.N. Fedorov", Kaluga
  - Federal State Autonomous Institution "Interdistrict Scientific and Technical Complex "Eye Microsurgery" named after Academician S.N. Fedorov" of the Ministry of Healthcare of the Russian Federation, Khabarovsk
  - "Angris", Limited Liability Company, Moscow
  - Moscow Medical university n.a. Sechenov, Moscow
  - Federal State Autonomous Institution "Interdistrict Scientific and Technical Complex "Eye Microsurgery" named after Academician S.N. Fedorov" of the Ministry of Healthcare of the Russian Federation, Moscow
  - Federal State Budgetary Educational Institution of Higher Education "Moscow State University of Medicine and Dentistry named after A.I. Evdokimov" of the Ministry of Healthcare of the Russian Federation, Moscow
  - "Moscow Regional Clinical Research Institute named after M.F. Vladimirsky", Moscow
  - Federal budgetary healthcare institution Privolzhsky district medical center FMBA of Russia., Nizhny Novgorod
  - Federal State Autonomous Institution "Interdistrict Scientific and Technical Complex "Eye Microsurgery" named after Academician S.N. Fedorov" of the Ministry of Healthcare of the Russian Federation, Novosibirsk
  - Budgetary Healthcare Institution of the Omsk Region "Clinical Eye Hospital named after V.P. Vykhodtsev, Omsk
  - Federal State Autonomous Institution "Interdistrict Scientific and Technical Complex "Eye Microsurgery" named after Academician S.N. Fedorov" of the Ministry of Healthcare of the Russian Federation, Saint Petersburg
  - "X7 Clinical Research", Limited Liability Company, Saint Petersburg
  - Feral State Budgetary Healthcare Institution "Clinical Hospital No. 122 named after L.G. Sokolov of the Federal Medical and Biological Agency", Saint Petersburg
  - Samara medical university, Samara
  - Nongovernmental Healthcare Institution "Clinical Hospital "RZhD [Russian Railways]-, Saratov
  - State Budgetary Institution "Ufa Research Institute of Eye Diseases of the Academy of Sciences of the Republic of Bashkortostan, Ufa
  - ZAO "Optimedservice", Ufa
  - Ulyanovsk ophthalmology clinical "Prozrenie", Ulyanovsk
  - Federal Budgetary Healthcare Institution "Volga Region Medical Centre" of the Federal Medical and Biological Agency, Veliky Novgorod
  - Federal State Autonomous Institution "Interdistrict Scientific and Technical Complex "Eye Microsurgery" named after Academician S.N. Fedorov" of the Ministry of Healthcare of the Russian Federation, Volgograd

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BRIN-20-01 | Azopt®
Started | 297 | 300
Completed | 287 | 289
Not Completed | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BRIN-20-01 | Azopt® | Total
Number analyzed (Participants) | 297 | 300 | 597
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (12.01) | 61.3 (12.01) | 61.2 (12.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170 | 174 | 344
  Male | 127 | 126 | 253
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 99 | 105 | 204
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 198 | 194 | 392
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Intraocular Pressure of Both Eyes Between the Two Treatment Groups
Description: The recommended primary endpoint is the mean difference in Intraocular Pressure of both eyes between the two treatment groups at pre-specified time points.
Time Frame: Baseline, Week 2 & Week 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | BRIN-20-01 | Azopt®
Number analyzed (Participants) | 273 | 271
mmHg
  Baseline- Left Eye 08:00 | 24.92 (2.290) | 25.06 (2.363)
  Baseline- Right Eye 08:00 | 24.87 (2.378) | 25.12 (2.358)
  Baseline - Left Eye 10:00 | 24.54 (2.307) | 24.83 (2.389)
  Baeline - Right Eye 10:00 | 24.52 (2.423) | 24.90 (2.365)
  Week 2 - Left Eye 08:00 | 19.87 (3.436) | 19.56 (3.642)
  Week 2 - Right Eye 08:00 | 19.81 (3.400) | 19.62 (3.423)
  Week 2 - Left Eye 10:00 | 18.87 (3.544) | 18.39 (3.760)
  Week 2 - Right Eye 10:00 | 18.69 (3.572) | 18.47 (3.468)
  Week 6 - Left Eye 08:00 | 18.86 (3.162) | 18.91 (3.333)
  Week 6 - Right Eye 08:00 | 18.87 (3.067) | 18.99 (3.123)
  Week 6 - Left Eye 10:00 | 17.76 (3.252) | 17.73 (3.418)
  Week 6 - Right Eye 10:00 | 17.71 (3.190) | 17.70 (3.162)
Statistical Analysis 1: Comparison: BRIN-20-01 vs Azopt®; Test type: Equivalence — Type of Statistical Test - Therapeutic equivalence. Sample size was based on 90% power at an alpha=0.05 significance level when the true difference between the means is 0 and SD=3.5 and the 95% equivalence limits are -1.0 and 1.0; 20% dropout was assumed; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [-0.28 to 0.91] — The reported mean difference represents value for Left Eye at Week 2, 08:00am
Statistical Analysis 2: Comparison: BRIN-20-01 vs Azopt®; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.39 to 0.76] — The reported mean difference represents value for Right Eye at Week 2, 08:00am
Statistical Analysis 3: Comparison: BRIN-20-01 vs Azopt®; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.59 to 0.50] — The reported mean difference represents value for Left Eye at Week 6, 08:00am
Statistical Analysis 4: Comparison: BRIN-20-01 vs Azopt®; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.64 to 0.40] — The reported mean difference represents value for Right Eye at Week 6, 08:00am

2. Secondary Outcome: Change From Baseline in IOP of Both Eyes Between the 2 Treatment Groups.
Time Frame: approximately 8:00 AM. (hour 0; before the morning drop) and 10:00 AM. (hour 2) at the Day 14 (Week 2) and Day 42 (Week 6) visits
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | BRIN-20-01 | Azopt®
Number analyzed (Participants) | 273 | 271
mmHg
  Week 2- Left Eye 08:00 | -4.67 (3.441) | -5.27 (3.617)
  Week 2- Right Eye 08:00 | -4.71 (3.286) | -5.28 (3.531)
  Week 2- Left Eye 10:00 | -5.68 (3.475) | -6.44 (3.717)
  Week 2 - Right Eye 10:00 | -5.82 (3.484) | -6.43 (3.630)
  Week 6- Left Eye 08:00 | -5.68 (3.290) | -5.92 (3.577)
  Week 6- Right Eye 08:00 | -5.64 (3.107) | -5.91 (3.468)
  Week 6 - Left Eye 10:00 | -6.78 (3.329) | -7.10 (3.614)
  Week 6 - Right Eye 10:00 | -6.81 (3.239) | -7.20 (3.500)
Statistical Analysis 1: Comparison: BRIN-20-01 vs Azopt®; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0015, two-sample t-test — P value reported for Left Eye at Week 2; 08:00 am
Statistical Analysis 2: Comparison: BRIN-20-01 vs Azopt®; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0008, two-sample t-test; P value reported for Right Eye at Week 2; 08:00am
Statistical Analysis 3: Comparison: BRIN-20-01 vs Azopt®; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < .0001, two-sample t-test; P value reported for left eye at week 6, 08:00 am
Statistical Analysis 4: Comparison: BRIN-20-01 vs Azopt®; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < .0001, two-sample t-test; P value reported for Right eye at Week 6; 08:00 am

ADVERSE EVENTS:
Time Frame: 7 Weeks
Arm/Group | BRIN-20-01 | Azopt®
All-Cause Mortality (participants affected / at risk) | 0/297 | 0/300
Serious Adverse Events (participants affected / at risk) | 0/297 | 1/300
Other Adverse Events (participants affected / at risk) | 49/297 | 38/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BRIN-20-01 (N=297) | Azopt® (N=300)
Hypertensive Crisis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BRIN-20-01 (N=297) | Azopt® (N=300)
Arrhythmia (Cardiac disorders) | 1 | 0
Abnormal Sensation in Eye (Eye disorders) | 1 | 0
Blepharitis (Eye disorders) | 1 | 1
Cataract (Eye disorders) | 1 | 0
Conjunctival Hyperemia (Eye disorders) | 3 | 2
Conjunctival Oedema (Eye disorders) | 0 | 1
Conjunctivitis Allergic (Eye disorders) | 0 | 2
Dry Eye (Eye disorders) | 2 | 0
Eye Irritation (Eye disorders) | 3 | 2
Eye Pain (Eye disorders) | 0 | 2
Eye Pruritus (Eye disorders) | 2 | 2
Foreign Body Sensation in Eyes (Eye disorders) | 4 | 2
Keratitis (Eye disorders) | 1 | 0
Lacrimation Increased (Eye disorders) | 1 | 0
Ocular Hyperemia (Eye disorders) | 3 | 2
Swelling of Eyelid (Eye disorders) | 1 | 0
Vision Blurred (Eye disorders) | 8 | 4
Visual Acuity Reduced (Eye disorders) | 0 | 1
Visual Impairment (Eye disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Instillation Site Dryness (General disorders) | 1 | 0
Instillation Site Pain (General disorders) | 2 | 0
Instillation Site Pruritus (General disorders) | 1 | 0
Instillation Site Reaction (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Respiratory Tract Infection Viral (Infections and infestations) | 1 | 2
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 1
Blood Pressure Increased (Investigations) | 2 | 1
Intraocular Pressure Increased (Investigations) | 0 | 1
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 6 | 8
Headache (Nervous system disorders) | 3 | 3
Breast Cyst (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertensive Crisis (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has exclusive rights, including the right of authorship, to all publications concerning Study data and findings. The Institution, the Investigator, and the Co-Investigators are contractually bound not to make any publications, public statements, oral presentations concerning the Study data and findings.

The Sponsor shall have the sole right to review, use, publish, and disclose any data, information, or results developed without limitation.

DOCUMENTS (2):
  • Study Protocol (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT05022004/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT05022004/SAP_001.pdf